CLINICAL TRIAL: NCT01677936
Title: A Randomized, Unblinded, Single Research Site, Comparator Study of Raisins Versus Alternative Snacks on Glycemic Control and Other Cardiovascular Risk Factors in Patients With Type 2 Diabetes Mellitus
Brief Title: Study of Raisins Versus Alternative Snacks in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Louisville Metabolic and Atherosclerosis Research Center (Other)
Collaborators: California Raisin Marketing Board (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Raisin DM 002
Record Dates: First submitted 2012-08-21; First posted 2012-09-03 (Estimated); Results first posted 2014-04-23 (Estimated); Last update posted 2014-04-23 (Estimated); Status verified 2014-03

CONDITIONS: Diabetes Mellitus
Keywords: diabetes; blood pressure; lipid; waist circumference; BMI
MeSH Terms: conditions — Diabetes Mellitus | interventions — Snacks

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Raisin (Experimental): Subjects randomized to the raisin treatment arm will consume raisins three times a day, prior to meals, and with a glass of water or non-caloric beverages (i.e. tea). Subjects will consume the raisins over a 12 week period.
  Interventions: Other: Raisins
- Snack Group (Active Comparator): Subjects randomized to the snack group will consume 100 calorie snack packs three times a day, before meals, and with water or other non-caloric beverages (i.e. tea). Subjects will consume the snack packs over a 12 week period.
  Interventions: Other: Snacks

INTERVENTIONS:
Other: Raisins — 1 oz, 90 calorie packages of raisins will be administered to subjects in the raisin treatment arm
  Arms: Raisin
Other: Snacks — 100 calorie snack packs will be administered to the subjects in the snack group
  Other Names: 100 calorie snack packs
  Arms: Snack Group

SUMMARY:
The objective of this study is to compare the effects of Raisins three times per day versus alternative snacks three times per day on blood sugar control and cardiovascular risk factors (weight, waist circumference, blood pressure, cholesterol levels) in patients with Type 2 Diabetes Mellitus. These effects will be studied over a 12 week period.

DETAILED DESCRIPTION:
Raisins are often considered a good food choice because they provide dietary fiber and many health-promoting nutrients, antioxidants and phytochemicals. Like most other fruits, raisins are devoid of fat, saturated fat and cholesterol, and low in sodium; these features, combined with their high potassium content, high fiber, and low glycemic index make them potentially preferable to other foods in their effects upon glycemic control and cardiovascular risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Are generally healthy men and women older than 18 years of age
* Are willing and able to undergo an informed consent process
* Have medical history of Type 2 Diabetes Mellitus
* Have hemoglobin A1c 67.5 - 10%
* Have body mass index (BMI) 25.0 to 39.9 kg/m2
* Have blood pressure > 100 mmHg systolic or > 70 mmHg diastolic
* Are willing and able to perform self-glucose monitoring throughout the study
* Are willing to fast before study visits
* Are willing and able to bring in their morning anti-diabetes mellitus drugs to study visits
* Women must be of non-childbearing potential defined as postmenopausal for at least 2 years or surgically sterile (i.e. bilateral tubal ligation, bilateral oophorectomy, or hysterectomy).
* If not menopausal or surgically sterile, then women of child-bearing potential must be willing to use:

  * oral contraceptives and another acceptable form of birth control, or
  * double barrier birth control methods such as condom or occlusive cap (e.g. diaphragm or cervical/vault caps) plus spermicidal agent (e.g. foam, gel, film, cream, suppository).
* Are willing to notify the research staff of any change in their medical health & concomitant medications/supplements during the course of the clinical trial

Exclusion Criteria:

* Intolerance, dislike, or unwillingness to consume raisins or any of the comparator snacks and affiliated ingredients
* History of greater than one drug allergy
* History of greater than one "food allergy"
* Change in anti-diabetes mellitus medication within 3 months prior to screening visit
* Change in blood pressure and/or lipid-altering medications within 1 month of screening visit
* Plans to change current anti-diabetes mellitus, blood pressure, or lipid-altering medications during course of the study
* Unwilling to maintain current anti-diabetes mellitus, blood pressure, or lipid-altering medications and their doses during the course of the study
* History of clinically significant diabetes mellitus complications, that in the opinion of the investigator, may interfere with the successful completion of the trial
* History of clinically significant diabetes mellitus kidney disease (e.g. clinically significant proteinuria)
* History of severe high or low blood sugars within the past year, as per Investigator discretion
* History of severe high or low blood sugars requiring hospitalization at any time in the past
* Subjects are excluded if within the past 6 months, they have history of myocardial infarction, acute coronary syndrome, stroke, or any cardiac / vascular surgical procedure (e.g. atherosclerotic coronary heart disease by-pass, carotid surgery, peripheral vascular by-pass, stent placement, pacemaker placement, etc.), unstable angina, or alterations in treatment of stable angina
* Subjects are excluded if at any time in the past, they have history of clinically significant ventricular or atrial dysrhythmias
* Subjects are excluded if at any time in the past, they have history of New York Heart Association (NYHA) functional heart failure of Class III or greater, defined as: CLASS III: Marked limitation of physical activity, comfortable at rest, but less than ordinary activity causes fatigue, palpitations or dyspnea, CLASS IV: Unable to carry out any physical activity without discomfort, symptoms of cardiac insufficiency at rest, if any physical activity is undertaken, discomfort is increased
* Subjects are excluded if at any time in the past, they have history of or known increases in QTc
* History of seizures in the past year
* Is pregnant, breastfeeding or plans to become pregnant during the course of the clinical trial
* Major surgical procedure within 30 days prior to visit #1 (i.e. day of signing of the informed consent document), or current plans to have a major surgical procedure during study participation or 30 days following completion of all study related procedures
* History of gastrointestinal malabsorption (e.g. uncontrolled crohn's disease, etc.) or history of a gastric bypass or other diversional bariatric surgery. Gastric banding procedure is also exclusionary if adjusted within 30 days prior to visit #1 (i.e. day of signing the informed consent document), or a reasonable chance of having a gastric banding adjustment during the course of the study
* History of ongoing malignancy. History of malignancy is acceptable for eligibility if successfully treated, with no evidence of persistence or recurrence of the malignancy within 5 years of visit #1 (i.e. day of signing the informed consent document) or basal carcinoma of the skin and "in situ" cancer of the cervix successfully treated 30 days prior to visit #1
* History of organ transplant.
* History of drug (licit or illicit) or alcohol abuse/addiction within 5 years of visit #1 (i.e. day of signing the informed consent document)
* Routinely consumes more than 2 units of alcohol per day. A unit of alcohol is defined as a 12 ounce (350 ml) beer, 5 ounce (150 ml) wine, or 1.5 ounce (45 ml) of 80-proof alcohol for mixed drinks.
* History of clinically significant heart, vascular, hematologic, orthopedic, rheumatologic, muscle, brain, neurologic (e.g. dementia, uncontrolled seizure disorder, etc.) , gastrointestinal (such as chronic hepatitis B or C, malabsorptive intestinal diseases such as uncontrolled crohn's disease, ulcerative colitis, severe irritable bowel syndrome, other significant gastrointestinal diseases that may interfere with study participation and/or results), endocrine (uncontrolled hyper or hypothyroidism), ophthalmologic, infectious (e.g. human immunodeficiency virus, tuberculosis, etc.) immunologic, nephrologic, pulmonary (e.g. poorly controlled asthma, poorly controlled chronic obstructive pulmonary disease, dyspnea, etc.), dermatologic, reproductive, psychiatric (e.g. bipolar disorder, schizophrenia, borderline personality disorder, etc.) disorders, or any other conditions that would present unacceptable risk to study subjects, compromise the acquisition or interpretation of study data, or otherwise interfere with the study subject's participation in the study.
* History of severe or uncontrolled depression based upon the opinion of the Principal Investigator.
* Blood pressure >160 mmHg systolic or >100 mmHg diastolic.
* Weight change (increase or decrease) of > 5 pounds in 2 months (by history) prior to visit 1
* Bradycardia defined as pulse less than 50 beats/minute
* History of clinically significant anemia
* Fasting serum lipoprotein values of: LDL-cholesterol, >160 mg/dl or triglycerides, >500 mg/dl (exclusionary during screening only)
* Creatinine level on screening > 1.5 times the upper range of normal.
* Liver enzymes on screening > 2 times the upper limits of normal
* Potassium level above the upper range of normal upon screening (one repeat lab would be permitted if the initial elevated potassium level is thought possibly due to laboratory error)
* Known laboratory abnormalities prior to randomization which Principal Investigator deems may pose an unacceptable risk, compromise acquisition or interpretation of study data, or otherwise interfere with the study subject's participation in the study
* Known positive testing for hepatitis B surface antigen, hepatitis C antibody, active hepatitis A immunoglobulin M, or human immunodeficiency virus (HIV)
* Current or past use of insulin
* Use of systemic corticosteroids (intravenous, subcutaneous, intra-articular). Inhaled and intranasal corticosteroids are permitted.
* Use of antiobesity/weight maintenance drug therapies at initial study visit, or within 2 months of the initial study visit.
* Use of digoxin or other cardiac antidysrhythmic drugs
* Use of anticoagulants (such as warfarin, Coumadin)
* Use of dietary supplements are acceptable, as long as the supplement intake was constant for one month prior to visit 1, and the study participant plans to continue the same supplement at the same dose throughout the study
* Known medical history of clinical significance, or any other conditions that would present unacceptable risk to study subject, compromise the acquisition or interpretation of study data, or otherwise interfere with the study subject's participation in the study as per discretion of the Principal Investigator.
* Is an employee or immediate family member of the research staff.
* Donated blood within 2 months prior to study entry, or plans to donate blood during the course of this study.
* Anticipation of a significant change in job, job duties, or job work hours, which might impair their ability and willingness to undergo study-related procedures under the timelines specified by protocol, and otherwise impede their completion of the study.
* Anticipation of or a reasonable likelihood of moving away from the research site, wherein such a move might impair their ability and willingness to undergo study-related procedures within the timelines specified by protocol, or otherwise impede their completion of the study.
* Anticipation of or a reasonable likelihood of vacations or other times away from home which might impair their ability and willingness to undergo study-related procedures within the timelines specified by the study protocol, or otherwise impede their completion of the study.
* Planned or anticipated major changes in lifestyle health practices, except as allowed by study protocol.
* Treatment with an investigational product or an investigational device within 30 days prior to visit #1 (i.e. day of signing the informed consent document) and have no plans to potentially start any investigational product or use an investigational device during or 30 days after the study subject completes all study related procedures.
* Reasonable life-expectancy of less than 2 years.
* Any other reason, if in the opinion of the Investigator, the individual study subject is not appropriate, or suitable for participation in the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2012-06; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harold E Bays, MD, Principal Investigator — L-MARC Research Center
Locations (1):
- L-MARC Research Center, Louisville, Kentucky, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 51 total subjects were randomized. 5 were excluded (1 snack; 4 raisin) due to lack of post-randomization evaluable data. Thus, the full analysis data set included 27 raisin and 19 snack.
Period: Overall Study
Arm/Group | Raisin | Snack Group
Started | 31 (31 randomized to raisins; 4 excluded due to lack of post-baseline evaluation; 27 = full dataset) | 20 (20 randomized to snacks; 1 excluded due to lack of post-baseline evaluation; 19 = full dataset)
Completed | 22 (Full analysis dataset completers) | 15 (Full analysis dataset completers)
Not Completed | 9 | 5
Not completed — Lost to Follow-up | 4 | 1
Not completed — Protocol Violation | 3 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 0 | 4

BASELINE CHARACTERISTICS:
Population: 51 total subjects were randomized. 5 were excluded (1 snack; 4 raisin) due to lack of post-randomization evaluable data. Thus, the full analysis data set included 27 raisin and 19 snack.
Groups:
- Total: Total of all reporting groups
Arm/Group | Raisin | Snack Group | Total
Number analyzed (Participants) | 27 | 19 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (8.56) | 59 (12.54) | 58 (10.22)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 10 | 31
  >=65 years | 6 | 9 | 15
Gender [Number; unit: participants]
  Female | 17 | 11 | 28
  Male | 14 | 9 | 23
Region of Enrollment [Number; unit: participants]
  United States | 27 | 19 | 46

OUTCOME MEASURES:

1. Primary Outcome: Postprandial Glucose Levels
Description: Raisins versus snacks: percent change in postprandial glucose levels at week 12
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Raisin | Snack Group
Number analyzed (Participants) | 22 | 16
percent | -6 (24) | 17 (36)
Statistical Analysis 1: Comparison: Raisin vs Snack Group; Test type: Superiority or Other; p = 0.024, t-test, 2 sided — Compared to snacks, raisins reduced percent post-prandial glucose levels by 23%, which met the a priori threshold for statistical significance; Mean Difference (Final Values) = 23

2. Secondary Outcome: Systolic Blood Pressure
Description: Raisins versus snacks: mmHg change in systolic blood pressure at week 12
Time Frame: 12 weeks.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Raisin | Snack Group
Number analyzed (Participants) | 27 | 19
mmHg | -4.2 (13) | 4.5 (14)
Statistical Analysis 1: Comparison: Raisin vs Snack Group; Test type: Superiority or Other; p = 0.035, t-test, 2 sided — Compared with snacks, the 8.8 mmHg reduction with raisins met the a priori threshold for statistical significance; Mean Difference (Final Values) = 8.7

ADVERSE EVENTS:
Groups:
- Raisin: Raisin group
- Snacks: Snack group
Arm/Group | Raisin | Snacks
Serious Adverse Events (participants affected / at risk) | 1/27 | 0/19
Other Adverse Events (participants affected / at risk) | 8/27 | 0/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Raisin (N=27) | Snacks (N=19)
Pulmonary embolus (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Regarding safety, only one Serious Adverse Experience occurred in a raisin administered subject who experienced a pulmonary embolus after a surgical procedure of hip replacement.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Raisin (N=27) | Snacks (N=19)
Gastrointestinal complaints (Gastrointestinal disorders) | 8 (8) | 0 (0) — Gastrointestinal complaints

LIMITATIONS AND CAVEATS:
This study was limited by being an un-blinded, single site study of modest size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No